CLINICAL TRIAL: NCT06446674
Title: Comparison Between Mini Monaka,Perforated Plugs and 3-Snip Punctoplasty in Punctal Stenosis.
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Almoatz bellah zohier Mohammed, Ophthalmology Specialist, Assiut University
Other Study IDs: PS
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Punctal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mini monaka — mini monaka,perforated plugs

SUMMARY:
To compare the result of mini monaka to perforated plug and 3 snip punctoplasty in management of punctal stenosis.

DETAILED DESCRIPTION:
Punctal stenosis is a common disorder of the punctum. It is an important cause of epiphora and accounted for 8% of all patients presenting with epiphora and 3% of all lacrimal drainage disorders. Although numerous factors have been implicated as causative agents, the exact pathogenesis is still elusive. The widely believed hypothesis that histological studies have supported is a common mechanism involving inflammation leading to fibrosis and subsequent stenosis .A stenotic punctum can be easily diagnosed by slit-lamp examination, while probing and irrigation of the lacrimal pathway is usually required to exclude a more distal obstruction There are no uniformly acceptable guidelines for the management of punctal stenosis. Several modalities described include punctal dilatation, 1-snip punctoplasty, 2-snip punctoplasty, 3-snip punctoplasty, rectangular 3-snip punctoplasty, 4-snip punctoplasty, punctal punching with Kelly's or Rsess punch, punctoplasty with mitomycin C, balloon punctoplasty, balloon puncta-canaliculoplasty, and inserting perforated punctal plugs, self-retaining bicanaliculata stents, or Mini-Monaka . The mini-monaka is a silicone post canalicular stent designed to repair canalicular lacerations. It is designed to fit snugly into the punctum and ampulla without any suturing .A perforated punctal plug can be put into the opening of the tear canal to allow drainage of tears. These are very small silicone arrowhead shaped tubes It is important to note that there is increasing evidence about the benefits of minimally invasive modalities like Mini-Monaka. the non-surgical dilation can be performed as an office procedure .

ELIGIBILITY:
Inclusion Criteria:

* o Confirmed unilateral or bilateral cases of punctal stenosis based on slit-lamp examination.

Exclusion Criteria:

* o Epiphora due to distal obstruction

  * Active ocular infection or inflammation.
  * Anatomic abnormalities
  * Ocular cicatricial pemphigoid

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be divided into 3 groups:
  Group A: 7 patients with punctal stenosis will be treated with mini monoka. Group B: 7 patients with punctal stenosis will be treated with punctoplasty. Group C: 7 patients with punctal stenosis will be treated with perforated plug
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Comparison between mini monaka,perforated plugs and 3-Snip punctoplasty in punctal stenosis by using slit lamp examination | 1 year
  correlation between mini monaka, perforated plugs and punctoplasty in punctal stenosis according to improvement in tear drainage by using slit lamp examination.
Comparison between mini monaka,perforated plugs and 3-Snip punctoplasty in punctal stenosis by using fluoresceine dilution test | 1 year
  correlation between mini monaka, perforated plugs and punctoplasty in punctal stenosis according to improvement in tear drainage by using fluoresceine dilution test

CONTACTS AND LOCATIONS:
Overall Officials: mohamed shehata, prof, Study Chair — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atkova EL, Maydanova AA, Krakhovetskiy NN, Reznikova LV. [Punctal stenosis: etiology, diagnosis, treatment]. Vestn Oftalmol. 2022;138(2):100-107. doi: 10.17116/oftalma2022138021100. Russian. PMID 35488568
- [Result] Bukhari AA. Management options of acquired punctal stenosis. Saudi Med J. 2013 Aug;34(8):785-92. PMID 23974448
- [Result] Tawfik HA, Ali MJ. A major review of punctal stenosis: Updated anatomy, epidemiology, etiology, and clinical presentation. Surv Ophthalmol. 2024 May-Jun;69(3):441-455. doi: 10.1016/j.survophthal.2024.02.001. Epub 2024 Feb 8. PMID 38336342
- [Result] Mansur C, Pfeiffer ML, Esmaeli B. Evaluation and Management of Chemotherapy-Induced Epiphora, Punctal and Canalicular Stenosis, and Nasolacrimal Duct Obstruction. Ophthalmic Plast Reconstr Surg. 2017 Jan/Feb;33(1):9-12. doi: 10.1097/IOP.0000000000000745. PMID 27429222
- [Result] Elbakary MA. Management of Bi-Punctal Stenosis by One-Snip Punctoplasty Combined with Silicone Intubation. Orbit. 2022 Jun;41(3):324-328. doi: 10.1080/01676830.2021.1904424. Epub 2021 Mar 29. PMID 33781149